CLINICAL TRIAL: NCT01409850
Title: Pilot Clinical Trial on the Treatment Effectiveness of Two Splints for Acute Temporomandibular Pain.
Brief Title: Comparison Study of Two Splints Used for Treatment of Acute Temporomandibular Pain.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very slow enrollment of participants
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Giannakopoulos Nikolaos, Dr.med.dent.,MSc, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UHeidelberg
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Myofascial Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aqualizer (Active Comparator)
  Interventions: Device: Aqualizer
- Soft splint (Active Comparator): elastic splint made of copolyester foil
  Interventions: Device: Soft splint
- Counselling (No Intervention)

INTERVENTIONS:
Device: Aqualizer — The Aqualizer is a soft splint with water-filled pads.
  Arms: Aqualizer
Device: Soft splint
  Arms: Soft splint

SUMMARY:
The most commonly applied treatment against acute temporomandibular signs and symptoms is pharmacotherapy. The evidence on treatment efficacy of non-medication treatments (like splints) is very low. Two very commonly used splints are the Aqualizer® and the soft polyester splint. These are splints applied for a short period of time, until the treatment with a hard splint and/or physiotherapy begins. Aim of this study is to compare the clinical short-time efficacy of these two splints for the treatment of acute temporomandibular pain and compare it to a control group receiving no therapy for that short time.

The study hypothesis is that there is a difference in pain reduction between the three groups of patients (two intervention and one control group).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, non-chronic orofacial pain

Exclusion Criteria:

* Pregnancy, chronic orofacial pain, dental treatment need, dental pain, edentulous space larger than 5mm, more than three molars missing in the same quadrant, rheumatic disease, Injury/operation in maxillofacial area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pain | 2-3 weeks

SECONDARY OUTCOMES:
mouth opening | 2-3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Prosthodontics, University Clinic of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany